CLINICAL TRIAL: NCT03327194
Title: Subjective Satisfaction and Audiological Benefit With ADHEAR Audio Processor and ADHEAR Adhesive Adapter in Children
Brief Title: Use of ADHEAR, a Non-Implantable Bone Conduction Hearing System, in Children With Single Sided Deafness and/or Conductive Hearing Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: MED-EL Elektromedizinische Geräte GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2017/ORL/ADHEAR
Record Dates: First submitted 2017-10-25; First posted 2017-10-31 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Conductive Hearing Loss; Single Sided Deafness
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Intervention Model Description: Monocentric prospective interventional single-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADHEAR Audio processor (Experimental)
  Interventions: Device: ADHEAR Audio Processor

INTERVENTIONS:
Device: ADHEAR Audio Processor — ADHEAR Audio Processoris a non-invasive bone conduction hearing device which is retained on the patient's head with an adhesive adapter that is placed behind the auricle.
  The ADHEAR Audio Processor transmits sounds to the mastoid by vibrating on the skull and stimulates the inner ear without any previous surgery.
  ADHEAR Audio Processor is classified as a Class lla medical device and ADHEAR Adhesive Adapter is classified as a Class I medical device.
  The ADHEAR Audio Processor has the CE mark.

SUMMARY:
A hearing loss affects the quality of life and the natural development of children.

The new generation of hearing devices provides a huge number of options to them. These new hearing aids are often aesthetically acceptable, less invasive and user-friendly.

The ADHEAR Non-Implantable Bone Conduction Hearing System is connected directly to the skin with a special adhesive adapter. The device transmits the sound to the mastoid by vibrating on the skull and stimulates the inner ear without any previous surgery.

The objective of this study is to evaluate of the audiological benefit and subjective satisfaction of ADHEAR Audio Processor with Adhesive attachment in a group of children suffering from conductive hearing loss and/or single sided deafness.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral and/or bilateral CHL (e. g. BC-thresholds <25dB HL)
* Ability to perform all tests required for the study
* Signed, and dated informed consent by parents and children where applicable

Exclusion Criteria:

* intolerant of the materials
* patient with a skin or scalp condition that may preclude the attachment of the adhesive plaster
* fluctuation of hearing loss over a two year period of 15dB in either direction
* retrocochlear, or central auditory disorders
* any physical, psychological, or emotional disorder that would interfere with the ability to perform on test and rehabilitation procedures

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximal decibels gain measured by Audiological basic tests | Week 3
Maximal decibels gain measured by speech reception threshold in quiet | Week 3

SECONDARY OUTCOMES:
Comparison of maximal decibels gain measured by Audiological basic tests between ADHEAR Audio Processor and Cochlear bone anchored hearing aid. | Day 0
Comparison of maximal decibels gain measured by speech reception threshold in quiet between ADHEAR Audio Processor and Cochlear bone anchored hearing aid | Day 0
Change from baseline in Quality of Life measured by the SSQ12 questionnaire | week 3
Change from baseline in Quality of Life measured by the SSQ12 questionnaire | month 3
Change from baseline in Quality of Life measured by the SSQ12 questionnaire | month 6
Change from baseline in Quality of Life measured by the SSQ12 questionnaire | month 12
Change from baseline in patient and parents satisfaction measured by the ADHEAR Questionnaire | week 3
Change from baseline in patient and parents satisfaction measured by the ADHEAR Questionnaire | month 3
Change from baseline in patient and parents satisfaction measured by the ADHEAR Questionnaire | month 6
Change from baseline in patient and parents satisfaction measured by the ADHEAR Questionnaire | month 12
Number of subjects who discontinue study device utilization due to any AE or dissatisfaction | Year 1
Average time of daily use of ADHEAR System | week 3
  Adherence reported by patient on a diary card.
Incidence of device-emergent adverse event. | Up to 1 year after start of study device utilization
  Number of participants with device-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Mansbach, MD PhD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Favoreel A, Heuninck E, Mansbach AL. Audiological benefit and subjective satisfaction of children with the ADHEAR audio processor and adhesive adapter. Int J Pediatr Otorhinolaryngol. 2020 Feb;129:109729. doi: 10.1016/j.ijporl.2019.109729. Epub 2019 Oct 15. PMID 31689608